CLINICAL TRIAL: NCT01851317
Title: The Relationship Between Patients' Position and Endotracheal Tube Intracuff Pressure in Pediatric Population
Brief Title: The Relationship Between Patients' Head Position and ETT Intracuff Pressure
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB13-00243
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Patients Undergoing ENT Surgery With Cuffed ETT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracuff pressure: Procedure/Surgery: Cuffed endotracheal tube

SUMMARY:
This study is designed to investigate the relationship between patients' position and endotracheal tube intracuff pressure in the pediatric population.

DETAILED DESCRIPTION:
There are currently no data in the literature as to the effect of changes in head position on CP. As the cuff is located in the patients' trachea, the shape of the patents' trachea may be change depending on the position of the patient's head and therefore, the CP may also change. If the intracuff pressure will increase as the patient's head is moved into a flexed or extended position, these patients may be at risk for tracheal damage. The investigators will prospectively evaluate the relationship between the patient's head position and CP in patients undergoing otolaryngological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 18 years
* Undergoing otolaryngological surgery with endotracheal intubation

Exclusion Criteria:

* Patient who is intubated with an uncuffed endotracheal tube
* Patients who have a limitation for movement of the neck or concerns of the stability of the cervical spine

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing otolaryngological surgery with cuffed endotracheal tube
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Endotracheal tube intracuff pressure | 1 day
  An intracuff pressure ≥ 30 cmH2O may compromise the tracheal mucosal perfusion and result in tracheal damage.

CONTACTS AND LOCATIONS:
Overall Officials: Hiromi Kako, M.D., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States